CLINICAL TRIAL: NCT06974929
Title: An Open-Label, Multicenter Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of HRS-6209 Combination Therapy in Patients With Breast Cancer
Brief Title: A Clinical Study of HRS-6209 Combined With Other Treatment Regimens in Patients With Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-6209-203
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-6209 in Combination with Letrozole Group (Experimental)
  Interventions: Drug: HRS-6209 Capsules; Drug: Letrozole Tablets
- HRS-6209 combined with Letrozole and HRS-2189 Group (Experimental)
  Interventions: Drug: HRS-6209 Capsules; Drug: Letrozole Tablets; Drug: HRS-2189 Tablets

INTERVENTIONS:
Drug: HRS-6209 Capsules — Oral HRS-6209 capsules.
Drug: Letrozole Tablets — Oral Letrozole tablets.
Drug: HRS-2189 Tablets — HRS-2189 tablets.
  Arms: HRS-6209 combined with Letrozole and HRS-2189 Group

SUMMARY:
This is a study to evaluate the safety, tolerability, and pharmacokinetic characteristics of HRS-6209 combined with other treatment regimens in breast cancer patients, and preliminarily observe its anti-tumor efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-75 years.
2. ECOG performance status 0-1.
3. Menopausal status.
4. Evidence of radiographic disease progression during or after the last systemic anti-tumor therapy prior to the first study drug administration.
5. At baseline, there must be at least one measurable, extracranial lesion that meets RECIST v1.1 criteria.
6. Expected survival > 3 months.
7. Women of childbearing potential must agree to use highly effective contraceptive measures during the study treatment and for 6 months after the end of treatment. Women of childbearing potential must have a negative serum HCG test within 7 days prior to study enrollment and must not be breastfeeding.
8. Voluntarily agree to participate in this clinical trial, willing and able to comply with the study visits and procedures, understand the study procedures, and have signed the informed consent form.

Exclusion Criteria:

1. Symptomatic visceral metastasis and other conditions, and the researcher judged that endocrine therapy was not suitable for use.
2. History of clinically serious cardiovascular disease.
3. The ECG examination was abnormal.
4. Patients with clinically significant endometrial abnormalities, including but not limited to endometrial hyperplasia and dysfunctional uterine bleeding.
5. The subjects were in acute infection or active tuberculosis and needed drug treatment.
6. The patients received surgery, chemotherapy, immunotherapy and macromolecular targeted therapy within 4 weeks before the first medication.
7. Pregnant and lactating women, or intending to become pregnant during the study.
8. There was a clear history of neurological or mental disorders and the subjects had a history of psychotropic drug abuse or drug abuse.
9. In the course of this study, it is expected to receive other anti-tumor treatments or drugs.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days after the first dose.
Maximum tolerated dose (MTD) | 28 days after the first dose.
Recommended phase II dose (RP2D) | 28 days after the first dose.
Adverse events (AEs) | About 1 year.
Serious adverse events (SAEs) | About 1 year.
Objective response rate (ORR) | About 1 year.

SECONDARY OUTCOMES:
Best overall response (BOR) | About 1 year.
Duration of response (DoR) | About 1 year.
Clinical benefit rate (CBR) | About 1 year.
Progression-free survival (PFS) | About 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided